CLINICAL TRIAL: NCT02434419
Title: Effect of Pectoral Electrostimulation on Reduction of Mammary Ptosis After Bariatric Surgery
Brief Title: Effect of Pectoral Electrostimulation on Reduction of Mammary Ptosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, MD, PhD, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HURJC2015-02
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PENS with training (Experimental): Patients undergoing percutaneous electrostimulation (PENS) of the pectoral muscle combined with specific training during 12 weeks postoperatively
  Interventions: Device: PENS; Other: Specific training
- Specific training (Active Comparator): Patients undergoing specific training during 12 weeks postoperatively
  Interventions: Other: Specific training
- No intervention (No Intervention): No specific treatment was assigned to these patients postoperatively

INTERVENTIONS:
Device: PENS — The participants underwent one 30-min session every week for 12 consecutive weeks. PENS was delivered by a needle electrode inserted in the medioclavicular line, 2 cm below the clavicle at a 90° angle towards the skin at a depth of approximately 1 cm. PENS was undertaken at frequency of 20 Hz at the highest amplify (0-20 mA) without causing pain. PENS was delivered simultaneously in both pectoral muscles.
  Arms: PENS with training
Other: Specific training — Patients underwent specific training exercises to improve pectoral fitness.
  Arms: PENS with training; Specific training

SUMMARY:
A prospective randomized clinical trial of patients undergoing bariatric surgery.

Patients were randomly assigned into 3 groups: those patients undergoing percutaneous electrostimulation (PENS) of the pectoral muscle combined with specific training (Group 1), those patients doing the specific training alone (Group 2) and those patients without any specific treatment (Group 3).

The assigned treatment began 15 days after surgery and was maintained during 12 weeks.

DETAILED DESCRIPTION:
A prospective randomized clinical trial of patients undergoing laparoscopic sleeve gastrectomy (LSG) or laparoscopic Roux-en-Y gastric bypass (RYGB) during 2014 was performed.

Patients were randomly assigned using a random-number table into 3 groups: those patients undergoing percutaneous electrostimulation (PENS) of the pectoral muscle combined with specific training (Group 1), those patients doing the specific training alone (Group 2) and those patients without any specific treatment (Group 3).

The assigned treatment began 15 days after surgery and was maintained during 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients with body mass index (BMI) >40 Kg/m2 or BMI > 35 Kg/m2 with the presence of comorbidities associated to obesity, undergoing a bariatric procedure.

Exclusion Criteria:

* all kind of previous breast surgery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Satisfaction degree. 7-points Likert scale was used for the quantification. | 12 weeks of treatment
  The patients were asked to quantify their satisfaction degree with the esthetic results of their breasts after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz-Tovar, MD, PhD, Principal Investigator — Hospital General Elche